CLINICAL TRIAL: NCT00771043
Title: Optical Coherence Tomography as a Measure of Neuroprotection in Patients With Relapsing-Remitting Multiple Sclerosis Receiving Natalizumab or Interferon Beta-1a
Brief Title: A Proof-of-Concept Study to Correlate Retinal Nerve Fiber Layer Changes in Patients With Multiple Sclerosis Treated With Natalizumab or Interferon Beta 1-a
Acronym: PRTOECT
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor decision to withdraw study at this time.
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: US 010-07-NAT
Record Dates: First submitted 2008-10-07; First posted 2008-10-10 (Estimated); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Relapsing-remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Natalizumab; Interferon beta-1a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TYSABRI (Experimental)
  Interventions: Drug: TYSABRI and AVONEX
- AVONEX (Experimental)
  Interventions: Drug: TYSABRI and AVONEX

INTERVENTIONS:
Drug: TYSABRI and AVONEX — TYSABRI and AVONEX treatment per package insert.

SUMMARY:
Phase IV, proof-of-concept, randomized, open-label, multi-center, two-arm, 9-month study to evaluate the neuroprotective effects of Natalizumab (TYSABRIÂ®) or Interferon beta-1a (AVONEXÂ®) treatments initiated at the time of acute optic neuritis (AON) as measured by RNFL thickness from Optical Coherence Tomography in patients with Relapsing Remitting Multiple Sclerosis (RRMS).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of RRMS.
* Patients with unilateral AON consistent with Multiple Sclerosis (MS).
* Treatment with intravenous methylprednisolone (IVMP) at 1gm daily for three days after the onset of AON, without a taper, and completed within 14 days of the AON symptom onset.
* Age 18-55 years.
* Expanded Disability Status Scale (EDSS) 0 to 5.0.
* Understand and sign informed consent.

Exclusion Criteria:

* History or presence of progressive multifocal leukoencephalopathy (PML).
* Diagnosis of Primary Progressive Multiple Sclerosis (PPMS) or Secondary Progressive Multiple Sclerosis (SPMS).
* Immune-compromised in the judgment of the Investigator.
* History of or presence of clinically significant medical illness or laboratory abnormality that, in the opinion of the investigator or Sponsor, would preclude participation in the study.
* Concomitant ophthalmologic disorders (e.g. diabetes, macular degeneration, etc).
* Previous history of severe disc edema, hemorrhage, or > 1 confirmed optic neuritis (ON) with the most recent ON symptom onset being less than 12 months ago.
* Previous treatment with > 1 Disease Modifying Therapy (DMT).
* Previous treatment with investigational products for MS, immunosuppressant or cytotoxic therapy.
* Previous treatment with TYSABRI®
* Women who are not postmenopausal, surgically sterile, or willing to practice contraception.
* Women pregnant, breast feeding, or planning to become pregnant.
* Involved with other study protocol simultaneously without prior approval.
* Determined not suitable for study participation by Investigator and/or Sponsor.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2008-11-01 (Actual); Primary Completion 2009-08-01 (Estimated); Study Completion 2010-06-01 (Estimated)

PRIMARY OUTCOMES:
Changes in average RNFL thickness as measured by OCT of affected eyes across treatment groups. | Between week 4 and weeks 36

SECONDARY OUTCOMES:
Changes in average RNFL thickness of affected eyes (corrected by fellow eyes) across treatment groups. | Between week 4 and weeks 36